CLINICAL TRIAL: NCT01226511
Title: A Double-Blind, Efficacy and Safety Study of Duloxetine Versus Placebo in the Treatment of Children and Adolescents With Generalized Anxiety Disorder
Brief Title: A Study in Pediatric Participants With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12929; F1J-MC-HMGI (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-12; First posted 2010-10-22 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Anxiety Neuroses; Anxiety States, Neurotic; Neuroses, Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): 30-120 mg flexible dosing once daily for 10 weeks. At the end of the 10 week blinded treatment period, participants may participate in an 18 week extension
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Administered once daily for 10 weeks. At the end of the 10 week blinded treatment period, placebo participants receive duloxetine in the 18 week extension
  Interventions: Drug: Duloxetine; Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: Cymbalta; LY248686
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out if duloxetine [30-120 milligrams (mg)] given once a day by mouth for 10 weeks to children and adolescents, is better than placebo when treating Generalized Anxiety Disorder (GAD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with GAD on clinical exam as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and supported by the Mini International Neuropsychiatric Interview for children and adolescents (MINI-Kid)
* Diagnosis of moderate or greater severity of GAD as determined by the following:

  * Presence of 4 or more symptoms identified on the generalized anxiety subsection of the Pediatric Anxiety Rating Scale (PARS) symptom checklist at screening and randomization. Two of which are excessive worry and dread or fearful anticipation (nonspecific)
  * PARS severity score of 15 or more at screening and randomization for symptoms identified on the generalized anxiety subsection of PARS symptom checklist at screening and randomization
  * Clinical Global Impressions of Severity (CGI-S) rating of 4 or more at screening and randomization
  * Presence of significant social, academic, and/or familial dysfunction as determined by the Children's Global Assessment Scale (CGAS) score of 60 or less at screening and randomization
* Female participants must test negative for pregnancy during screening Furthermore, female participants must agree to abstain from sexual activity or to use a reliable method of birth control as determined by the investigator during the study
* Participant's parent/legal representative and participant, if capable, are judged to be reliable by the investigator to keep all appointments for clinical visits, tests, and procedures required by the protocol
* Participant's parent/legal representative and participant, if capable, must have a degree of understanding such that they can communicate intelligently with the investigator and study coordinator
* Participants must be capable of swallowing study drug whole (without opening the capsule, crushing, dissolving, dividing, et cetera)
* Participants must have venous access sufficient to allow blood sampling and are compliant with blood draws as per the protocol

Exclusion Criteria:

* Current diagnosis of major depressive disorder (MDD)
* Participants for whom the primary focus of treatment is separation anxiety or social phobia (participants with secondary separation anxiety or social phobia are allowed to participate)
* Have current primary diagnosis of any DSM-IV-TR Axis I disorder except GAD, or a current secondary DSM-IV-TR Axis 1 disorder that requires any pharmacologic treatment (other than those disorders listed below). Primary is defined as the disorder that is the primary focus of treatment
* Have a history of DSM-IV-TR-defined substance abuse or dependence within the past year, excluding caffeine and nicotine
* Have a current or previous diagnosis of bipolar disorder, psychotic depression, schizophrenia or other psychotic disorder, anorexia, bulimia, obsessive compulsive disorder, post-traumatic stress disorder, panic disorder, or pervasive development disorder, as judged by the investigator
* Have 1 or more first-degree relatives (parents or siblings) with diagnosed bipolar I disorder
* Have a serious or unstable medical illness, psychological condition, clinically significant laboratory or electrocardiogram (ECG) result, hypersensitivity to duloxetine, or its active ingredients, frequent or severe allergic reactions to multiple medications, uncontrolled narrow-angle glaucoma, acute liver injury (for example, hepatitis) or severe cirrhosis (Child-Pugh Class C), or a history of any seizure disorder (other than febrile seizures)
* Have a significant suicide attempt within 1 year of screening or are currently at risk of suicide in the opinion of the investigator
* Have initiated, stopped, or changed the type or intensity of psychotherapy within 6 weeks prior to screening. Participants who require a change to psychotherapy between weeks 1 through 10 will be excluded
* Have a weight less than 20 kilograms at any time during the screening period
* Female participants who are pregnant, nursing or have recently given birth

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 281 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hialeah, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smyrna, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gladstone, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Insurgentes Cuicuilco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zona Centro
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria

REFERENCES:
- [Derived] Strawn JR, Prakash A, Zhang Q, Pangallo BA, Stroud CE, Cai N, Findling RL. A randomized, placebo-controlled study of duloxetine for the treatment of children and adolescents with generalized anxiety disorder. J Am Acad Child Adolesc Psychiatry. 2015 Apr;54(4):283-93. doi: 10.1016/j.jaac.2015.01.008. Epub 2015 Jan 29. PMID 25791145

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had 4 periods: Screening period (1-week), acute treatment period (10-week, double-blind period with flexible duloxetine dosing), extension treatment (18-week period, of which 16 weeks were open-label treatment with flexible duloxetine dosing), and a taper period (2 weeks recommended at discontinuation from study any point after Week 2).
Groups:
- Duloxetine/Duloxetine: Participants received flexible doses of duloxetine 30 to 120 milligrams (mg) orally, once daily (QD) for 10 weeks during the acute treatment period and flexible doses of duloxetine 30 to 120 mg orally, QD for 18 weeks during the optional extension treatment period. Duloxetine was provided in 30-mg capsules.
  Participants who received higher doses of duloxetine at the end of treatment period participation received gradually lower doses of duloxetine over the 2-week recommended tapering period, and participants who received the lowest dose of duloxetine or placebo at the end of treatment period participation received placebo over the 2-week recommended tapering period.
- Placebo/Duloxetine: Participants received placebo capsules orally, QD for 10 weeks during the acute treatment period and flexible doses of duloxetine 30 to 120 mg orally, QD for 18 weeks during the optional extension treatment period. Duloxetine was provided in 30-mg capsules.
  Participants who received higher doses of duloxetine at the end of treatment period participation received gradually lower doses of duloxetine over the 2-week recommended tapering period, and participants who received the lowest dose of duloxetine or placebo at the end of treatment period participation received placebo over the 2-week recommended tapering period.
Period: Acute Treatment Period
Arm/Group | Duloxetine/Duloxetine | Placebo/Duloxetine
Started | 140 (Thirty-one (31) participants who discontinued acute treatment did not enter the taper period.) | 141 (Twenty-six (26) participants who discontinued acute treatment did not enter the taper period.)
Completed | 108 | 110
Not Completed | 32 | 31
Not completed — Adverse Event | 7 | 6
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 3 | 6
Not completed — Parent/caregiver decision | 5 | 7
Not completed — Protocol Violation | 5 | 5
Not completed — Withdrawal by Subject | 10 | 6
Period: Extension Treatment Period
Arm/Group | Duloxetine/Duloxetine | Placebo/Duloxetine
Started | 108 (Nineteen (19) participants who discontinued extension treatment did not enter the taper period.) | 110 (Twenty-three (23) participants who discontinued extension treatment did not enter the taper period.)
Completed | 81 (Thirty-nine (39) participants who completed extension treatment did not enter the taper period.) | 83 (Thirty-five (35) participants who completed extension treatment did not enter the taper period.)
Not Completed | 27 | 27
Not completed — Adverse Event | 8 | 8
Not completed — Lack of Efficacy | 3 | 2
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Parent/Caregiver Decision | 8 | 8
Not completed — Sponsor Decision | 1 | 1
Period: Taper Period
Arm/Group | Duloxetine/Duloxetine | Placebo/Duloxetine
Started | 51 | 57
Completed | 46 | 54
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Parent/Caregiver Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants, excluding 9 participants from 1 site with major quality issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine/Duloxetine | Placebo/Duloxetine | Total
Number analyzed (Participants) | 135 | 137 | 272
Age, Customized [Number; unit: participants]
  7 to 11 years | 62 | 66 | 128
  12 to 17 years | 73 | 71 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 75 | 145
  Male | 65 | 62 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 40 | 77
  Not Hispanic or Latino | 88 | 88 | 176
  Unknown or Not Reported | 10 | 9 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 7 | 6 | 13
  Asian | 1 | 1 | 2
  Black or African American | 9 | 10 | 19
  White | 112 | 111 | 223
  More than 1 race | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 98 | 99 | 197
  Mexico | 26 | 26 | 52
  South Africa | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 10-Week Endpoint in the Pediatric Anxiety Rating Scale (PARS) Severity Score Evaluated for Symptoms Identified on the Generalized Anxiety Subsection of the PARS Symptom Checklist
Description: PARS severity score for GAD was assessed for all symptoms identified in the generalized anxiety section of the PARS symptom checklist. PARS severity score for GAD was derived by summing 5 of 7 severity/impairment/interference items (2, 3, 5, 6, 7); each item ranged from 0 (none) to 5 (extreme severity/impairment/interference). PARS severity scores for GAD ranged from 0 (none) to 25 (extreme severity), with a score of 15 indicating moderate illness severity. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach adjusted for baseline, pooled investigator, age category, visit, treatment, treatment*visit, age category*visit, and baseline*visit.
Time Frame: Baseline, 10 weeks
Population: Randomized participants with a baseline and at least 1 post-baseline PARS severity score for GAD during the acute treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine (Acute Treatment): Participants received flexible doses of duloxetine 30 to 120 milligrams (mg) orally, once daily (QD) for 10 weeks during the acute treatment period.
- Placebo (Acute Treatment): Participants received placebo capsules orally, QD for 10 weeks during the acute treatment period.
Arm/Group | Duloxetine (Acute Treatment) | Placebo (Acute Treatment)
Number analyzed (Participants) | 135 | 133
units on a scale | -9.70 (0.502) | -7.05 (0.500)
Statistical Analysis 1: Comparison: Duloxetine (Acute Treatment) vs Placebo (Acute Treatment); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Least squares (LS) mean difference = -2.65, 95% CI 2-sided [-4.03 to -1.27], Standard Error of Mean 0.700

2. Secondary Outcome: Response Rate at Endpoint for Generalized Anxiety Disorder (GAD) Using Pediatric Anxiety Rating Scale (PARS) Severity Score for GAD
Description: Response rate was defined as the percentage of participants having a 50% improvement from baseline to endpoint on the PARS severity score for GAD. PARS severity score for GAD was assessed for all symptoms identified in the generalized anxiety section of the PARS symptom checklist. PARS severity score for GAD was derived by summing 5 of 7 severity/impairment/interference items (2, 3, 5, 6, 7); each item ranged from 0 (none) to 5 (extreme severity/impairment/interference). PARS severity scores for GAD ranged from 0 (none) to 25 (extreme severity), with a score of 15 indicating moderate illness severity.
Time Frame: Baseline, 10 weeks
Population: Randomized participants with a baseline and at least 1 post-baseline PARS severity score for GAD [last observation carried forward (LOCF)] during the acute treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine (Acute Treatment) | Placebo (Acute Treatment)
Number analyzed (Participants) | 135 | 133
percentage of participants | 51 (4.8) | 37 (4.8)

3. Secondary Outcome: Change From Baseline to 10-Week Endpoint on the Pediatric Anxiety Rating Scale (PARS) Severity Total Score Evaluated for All Symptoms Identified on the PARS Symptom Checklist Symptoms
Description: PARS severity total score was assessed for all symptoms identified on the PARS symptom checklist. PARS severity total score was derived by summing 5 of 7 severity/impairment/interference items (2, 3, 5, 6, 7); each item ranged from 0 (none) to 5 (extreme severity/impairment/interference). PARS severity total scores ranged from 0 (none) to 25 (extreme severity), with a score of 15 indicating moderate illness severity. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach adjusted for treatment, pooled investigator, visit, baseline, age category, treatment*visit, baseline*visit, and age category*visit.
Time Frame: Baseline, 10 weeks
Population: Randomized participants with a baseline and at least 1 post-baseline PARS severity total score during the acute treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine (Acute Treatment) | Placebo (Acute Treatment)
Number analyzed (Participants) | 135 | 133
units on a scale | -9.15 (0.479) | -6.36 (0.477)

4. Secondary Outcome: Change From Baseline to 10-Week Endpoint on the Clinical Global Impression of Severity (CGI-S) Scale
Description: The CGI-S scale evaluated the severity of illness at the time of assessment. Scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill). Higher scores indicated a greater severity of illness. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach adjusted for treatment, pooled investigator, visit, baseline, age category, treatment*visit, baseline*visit, and age category*visit.
Time Frame: Baseline, 10 weeks
Population: Randomized participants with a baseline and at least 1 post-baseline CGI-S score during the acute treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine (Acute Treatment) | Placebo (Acute Treatment)
Number analyzed (Participants) | 135 | 133
units on a scale | -1.93 (0.114) | -1.38 (0.113)

5. Secondary Outcome: Remission Rate at Endpoint for Generalized Anxiety Disorder (GAD) Using Clinical Global Impressions of Severity (CGI-S) Scale
Description: Remission rate was defined as the percentage of participants having a CGI-S score ≤2 at endpoint. The CGI-S scale evaluated the severity of illness at the time of assessment. Scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill). Higher scores indicated a greater severity of illness.
Time Frame: 10 weeks
Population: Randomized participants with at least 1 post-baseline CGI-S score [last observation carried forward (LOCF)] during the acute treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine (Acute Treatment) | Placebo (Acute Treatment)
Number analyzed (Participants) | 135 | 133
percentage of participants | 45 | 30

6. Secondary Outcome: Change From Baseline to 10-Week Endpoint in the Children's Global Assessment Scale (CGAS)
Description: The CGAS was a clinician-rated assessment of general functioning. CGAS raw scores ranged from 1 (greatest impairment) to 100 (superior functioning). Lower scores indicated a lower level of functioning and greater impairment. Least squares (LS) mean from an analysis of covariance (ANCOVA) was adjusted for treatment, pooled investigator, baseline, and age category.
Time Frame: Baseline, 10 weeks
Population: Randomized participants with a baseline and at least 1 post-baseline [last observation carried forward (LOCF)] CGAS score during the acute treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine (Acute Treatment) | Placebo (Acute Treatment)
Number analyzed (Participants) | 123 | 124
units on a scale | 17.14 (1.232) | 12.16 (1.219)

7. Secondary Outcome: Percentage of Participants During the 10-Week Period With Treatment-Emergent (New or Worsening) Suicidal Ideation as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captured occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any 1 of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Results reported as percentage of participants with treatment-emergent (new or worsening) suicidal ideation from baseline=(number of participants with changes compared to baseline/total number of participants at risk)*100.
Time Frame: Baseline up to 10 weeks
Population: Randomized participants with a baseline and at least 1 post-baseline C-SSRS suicidal ideation score during the acute treatment period, whose baseline maximum C-SSRS suicidal ideation score was <5. Nine (9) participants from 1 site with major quality issues were excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine (Acute Treatment) | Placebo (Acute Treatment)
Number analyzed (Participants) | 135 | 134
percentage of participants | 5.9 | 5.2

8. Secondary Outcome: Percentage of Participants During the 10-Week Period With Treatment-Emergent (New or Worsening) Suicidal Behavior as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captured occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Reported as percentage of participants with treatment-emergent (new or worsening) suicidal behavior from baseline=(number of participants with changes compared to baseline/total number of participants at risk)*100.
Time Frame: Baseline up to 10 weeks
Population: Randomized participants with a baseline and at least 1 post-baseline C-SSRS suicidal behavior score during the acute treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine (Acute Treatment) | Placebo (Acute Treatment)
Number analyzed (Participants) | 135 | 134
percentage of participants | 0.0 | 0.0

9. Secondary Outcome: Change From 10-Week to 28-Week Endpoint in the Pediatric Anxiety Rating Scale (PARS) Severity Score Evaluated for Symptoms Identified on the Generalized Anxiety Subsection of the PARS Symptom Checklist
Description: PARS severity score for GAD was assessed for all symptoms identified in the generalized anxiety section of the PARS symptom checklist. PARS severity score for GAD was derived by summing 5 of 7 severity/impairment/interference items (2, 3, 5, 6, 7); each item ranged from 0 (none) to 5 (extreme severity/impairment/interference). PARS severity scores for GAD ranged from 0 (none) to 25 (extreme severity), with a score of 15 indicating moderate illness severity. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach adjusted for pooled investigator, visit, baseline, age category, baseline*visit, and age category*visit within reporting groups.
Time Frame: 10 weeks, 28 weeks
Population: Randomized participants with a PARS severity score for GAD during the acute treatment period and at least 1 PARS severity score for GAD during the extension treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine/Duloxetine (Extension Treatment): Participants received flexible doses of duloxetine 30 to 120 milligrams (mg) orally, once daily (QD) for 10 weeks during the acute treatment period and flexible doses of duloxetine 30 to 120 mg orally, QD for 18 weeks during the optional extension treatment period.
- Placebo/Duloxetine (Extension Treatment): Participants received placebo capsules orally, QD for 10 weeks during the acute treatment period and flexible doses of duloxetine 30 to 120 mg orally, QD for 18 weeks during the optional extension treatment period.
Arm/Group | Duloxetine/Duloxetine (Extension Treatment) | Placebo/Duloxetine (Extension Treatment)
Number analyzed (Participants) | 104 | 105
units on a scale | -3.33 (0.352) | -5.15 (0.452)

10. Secondary Outcome: Change From 10-Week to 28-Week Endpoint on the Pediatric Anxiety Rating Scale (PARS) Severity Total Score Evaluated for All Symptoms Identified on the PARS Symptom Checklist Symptoms
Description: PARS severity total score was assessed for all symptoms identified on the PARS symptom checklist. PARS severity total score was derived by summing 5 of 7 severity/impairment/interference items (2, 3, 5, 6, 7); each item ranged from 0 (none) to 5 (extreme severity/impairment/interference). PARS severity total scores ranged from 0 (none) to 25 (extreme severity), with a score of 15 indicating moderate illness severity. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach adjusted for pooled investigator, visit, baseline, age category, baseline*visit, and age category*visit within reporting groups.
Time Frame: 10 weeks, 28 weeks
Population: Randomized participants with a PARS severity total score during the acute treatment period and at least 1 PARS severity total score during the extension treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine (Extension Treatment) | Placebo/Duloxetine (Extension Treatment)
Number analyzed (Participants) | 104 | 105
units on a scale | -3.32 (0.357) | -5.26 (0.432)

11. Secondary Outcome: Change From 10-Week to 28-Week Endpoint on the Clinical Global Impression of Severity (CGI-S) Scale
Description: The CGI-S scale evaluated the severity of mental illness at the time of assessment. Scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill). Higher scores indicated a greater severity of illness. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach adjusted for pooled investigator, visit, baseline, age category, baseline*visit, and age category*visit within reporting groups.
Time Frame: 10 weeks, 28 weeks
Population: Randomized participants with a CGI-S score during the acute treatment period and at least 1 CGI-S score during the extension treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine (Extension Treatment) | Placebo/Duloxetine (Extension Treatment)
Number analyzed (Participants) | 104 | 105
units on a scale | -0.76 (0.093) | -1.17 (0.088)

12. Secondary Outcome: Change From 10-Week to 28-Week Endpoint in the Children's Global Assessment Scale (CGAS)
Description: The CGAS was a clinician-rated assessment of general functioning. CGAS raw scores ranged from 1 (greatest impairment) to 100 (superior functioning). Lower scores indicated a lower level of functioning and greater impairment. Least squares (LS) mean from an analysis of covariance (ANCOVA) was adjusted for pooled investigator, baseline, and age category within reporting groups.
Time Frame: 10 weeks, 28 weeks
Population: Randomized participants with a CGAS score during the acute treatment period and at least 1 CGAS score during the extension treatment period [last observation carried forward (LOCF)], excluding 9 participants from 1 site with major quality issues.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine (Extension Treatment) | Placebo/Duloxetine (Extension Treatment)
Number analyzed (Participants) | 103 | 105
units on a scale | 7.32 (1.19) | 10.48 (1.03)

13. Secondary Outcome: Percentage of Participants During the 18-Week Extension Period With Treatment-Emergent (New or Worsening) Suicidal Ideation as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: as for outcome 7
Time Frame: 10 weeks up to 28 weeks
Population: Randomized participants with a C-SSRS suicidal ideation score <5 at the last 2 visits in the acute treatment period and at least 1 C-SSRS suicidal ideation score during the extension treatment period. Nine (9) participants from 1 site with major quality issues were excluded.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine/Duloxetine (Extension Treatment) | Placebo/Duloxetine (Extension Treatment)
Number analyzed (Participants) | 104 | 105
percentage of participants | 3 | 3

14. Secondary Outcome: Percentage of Participants During the 18-Week Extension Period With Treatment-Emergent (New or Worsening) Suicidal Behavior as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: as for outcome 8
Time Frame: 10 weeks up to 28 weeks
Population: Randomized participants with a C-SSRS suicidal behavior score at the last 2 visits in the acute treatment period and at least 1 C-SSRS suicidal behavior score during the extension treatment period, excluding 9 participants from 1 site with major quality issues.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine/Duloxetine (Extension Treatment) | Placebo/Duloxetine (Extension Treatment)
Number analyzed (Participants) | 104 | 105
percentage of participants | 0 | 2

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were reported for all randomized participants, excluding 9 participants from 1 site with major quality issues.
Groups:
- Duloxetine: Adverse events (AEs) during the acute treatment period for participants who received flexible doses of duloxetine 30 to 120 milligrams (mg) orally, once daily (QD) for 10 weeks.
- Placebo: AEs during the acute treatment period for participants who received placebo capsules orally, QD for 10 weeks.
- Duloxetine/Duloxetine-Extension Treatment: AEs during the extension treatment period for participants who received flexible doses of duloxetine 30 to 120 mg orally, QD during both the acute and extension treatment periods (up to 28 weeks).
- Placebo/Duloxetine-Extension Treatment: AEs during the extension treatment period for participants who received placebo capsules orally, QD during the acute treatment period (10 weeks) and flexible doses of duloxetine 30 to 120 mg orally, QD during the extension treatment period (up to 18 weeks).
- Duloxetine-Taper: AEs during the taper period for participants who were dispensed duloxetine prior to entering the taper phase. Participants who received higher doses of duloxetine at the end of treatment period participation received gradually lower doses of duloxetine over the 2-week recommended tapering period.
- Placebo-Taper: AEs during the taper period for participants who were dispensed placebo prior to entering the taper phase. Participants who received the lowest dose of duloxetine or placebo at the end of treatment period participation received placebo over the 2-week recommended tapering period.
Arm/Group | Duloxetine | Placebo | Duloxetine/Duloxetine-Extension Treatment | Placebo/Duloxetine-Extension Treatment | Duloxetine-Taper | Placebo-Taper
Serious Adverse Events (participants affected / at risk) | 1/135 | 0/137 | 2/104 | 2/106 | 1/97 | 1/7
Other Adverse Events (participants affected / at risk) | 106/135 | 90/137 | 73/104 | 73/106 | 12/97 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=135) | Placebo (N=137) | Duloxetine/Duloxetine-Extension Treatment (N=104) | Placebo/Duloxetine-Extension Treatment (N=106) | Duloxetine-Taper (N=97) | Placebo-Taper (N=7)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — SAE reported for 1 participant (Duloxetine/Duloxetine group) during the extension treatment period and resolved during the duloxetine-taper period. The SAE was counted in both periods, although it was not new or worsening during the taper period.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine (N=135) | Placebo (N=137) | Duloxetine/Duloxetine-Extension Treatment (N=104) | Placebo/Duloxetine-Extension Treatment (N=106) | Duloxetine-Taper (N=97) | Placebo-Taper (N=7)
Palpitations (Cardiac disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 13 (15) | 9 (10) | 5 (6) | 7 (7) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 6 (6) | 1 (3) | 5 (6) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 28 (35) | 8 (8) | 10 (10) | 13 (16) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 22 (23) | 10 (10) | 5 (7) | 6 (6) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 11 (11) | 6 (6) | 4 (4) | 9 (9) | 0 (0) | 0 (0)
Irritability (General disorders) | 4 (4) | 6 (6) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (5) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 6 (6) | 4 (4) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 12 (13) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 6 (6) | 5 (5) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 20 (21) | 7 (7) | 1 (1) | 9 (10) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 10 (10) | 2 (2) | 5 (5) | 7 (9) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 27 (37) | 23 (29) | 13 (17) | 11 (13) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 16 (16) | 9 (9) | 3 (4) | 8 (11) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 12 (13) | 7 (8) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2/70 (3) | 2/75 (2) | 0/53 (0) | 2/59 (2) | 0/47 (0) | 0/3 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 3 (3) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Nine (9) randomized participants (5 duloxetine, 4 placebo) from 1 site were excluded from efficacy and safety analyses due to major quality issues at that site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days